CLINICAL TRIAL: NCT02739477
Title: Tolerance and Activity Assessment of High Doses of Favipiravir in Male Survivors With Ebola Virus in the Semen
Brief Title: Tolerance and Activity Evaluation of High Doses of Favipiravir Against Ebola Virus in the Semen
Acronym: FORCE
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: End date of epidemic
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C15-101
Record Dates: First submitted 2016-02-24; First posted 2016-04-15 (Estimated); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Ebola Virus Survivor
Keywords: Favipiravir; Tolerance; Survivor; Ebola Virus; Genital reservoir; Guinea
MeSH Terms: interventions — favipiravir

ARMS (1):
- Favipiravir (Experimental): Favipiravir (oral administration, 200 mg light yellow, round-shaped, coated divisible tablets that can be crushed and mixed with liquid)
  Interventions: Drug: Favipiravir

INTERVENTIONS:
Drug: Favipiravir — Cohort 1: Day 1 (inclusion) 4800 mg (2400 mg bid). Day 2 to Day 14: 3600 mg (1800 mg bid).
  Cohort 2: Day 1 (inclusion) 4800 mg (2400 mg bid). Day 2 to Day 14: 3600, 4200, 4800 mg per day depending on cohort 1 results.
  Cohort 3: Day 1 (inclusion) 4800 mg (2400 mg bid). Day 2 to Day 14: 3600, 4200, 4800 mg per day depending on cohorts 1 and 2 results.
  Other Names: AVIGAN

SUMMARY:
This study aims to evaluate favipiravir high dose tolerance in male survivor of Ebola Virus Disease (EVD) with Ebola Virus (EBOV) RNA in semen. This is a dose escalation study with 3 cohorts of 6 patients, each dose level including 2 sentinel patients.

DETAILED DESCRIPTION:
Rational:

* Data suggesting persistence of EBOV in semen a few months after the end of EVD and sexual transmission of EBOV
* Encouraging results on favipiravir efficacy to reduce mortality of EVD in JIKI trial (NCT02329054 )
* Favipiravir trough plasma concentration in JIKI trial lower than predicted by population pharmacokinetic model, suggesting an increase of dose might be necessary to achieve a therapeutically relevant exposure.

Objectives:

* Primary objective: to assess clinical and biological tolerance of high-dosed favipiravir bid for 14 days
* Secondary objectives: to assess the activity of favipiravir on evolution of EBOV RNA and infectious loads in semen under treatment; the trough plasma and semen concentrations of favipiravir; and genetic factors associated with favipiravir pharmacokinetic.

Dose escalation scheme:

Each patient of each cohort will receive favipiravir loading doses of 4800 mg at Day 1 (2400 mg bid), following by 3600 mg (1800 mg bid) from Day 2 to 14 (cohort 1), then 3600, 4200 or 4800 mg from Day 2 to 14 (cohort 2 and 3), depending on previous cohort results.

Escalation rules are based on the number of patient undergoing treatment-related adverse events (TRAE) of grade 3 or 4 according to the Common Terminology Criteria for Adverse Events v4.03 (CTCAE), as defined by the investigator and sponsor.

Participants will attend medical visits at Day 1, Day 3, Day 7, Day 10, Day 14, Day 21 and clinical tolerance will be assessed daily by phone call from Day 1 to Day 14.

At the end of the first cohort:

* if no TRAE, cohort 2 will be given 2400 mg bid from Day 2 to 14;
* if 1 or 2 TRAE is observed, cohort 2 will be given 2100 mg bid from Day 2 to Day 14;
* if 3 or more TRAE is observed, cohort 2 will be given the same dose as cohort 1.

At the end of cohort 2, same rules will be apply to cohort 3, without exceed 4800 mg of favipiravir per day.

Each cohort will include 6 patients. Each dose level will comprise 2 sentinel patients.

In their own interest, patients included in a cohort with detection of EBOV RNA in semen by RT-PCR (CT<38) at Day 21, could be included in the next cohort.

Recruitment will start among PostEbogui cohort from coast Guinea.

ELIGIBILITY:
Inclusion Criteria:

* male survivor of biologically confirmed EVD
* age >= 18 years
* EBOV RT-PCR on semen with cycle threshold [Ct]<38 at Day -7 and semen aliquot available for later quantification of EBOV
* signed informed consent

Non-Inclusion Criteria:

* EBOV RT-PCR on blood with cycle threshold [Ct]<38 at Day -7
* Biological abnormality higher than grade 2 according to CTCAE (v4.03) on following parameters: creatinine, ASAT, ALAT, alkaline phosphatase, total bilirubin
* Fridericia corrected QT interval (QTc) > 450 ms
* Concomitant use of QT/QTc interval-prolonging drugs or drugs that could cause electrolyte imbalance, such as: loop diuretics, thiazide diuretics or related
* Previous gout attack or ongoing treatment for gout or hyperuricemia
* Ongoing pyrazinamide treatment or other drug known to induce hyperuricemia
* Previous hypersensitivity reaction due to nucleoside analogue
* Symptom or biological value suggesting systemic disorder (renal, hepatic, cardio-vascular, pulmonary) or any medical condition that could interfere with results interpretation or compromise participants' health
* Explicit refusal to comply with proper use of drug (condom use)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2016-04; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Number of patients undergoing grade 3 or 4 clinical or biological adverse events related to Favipiravir (Common Terminology Criteria for Adverse Events, CTCAE, v4.03) | Day 14
  Day 1 is the first day of favipiravir intake

SECONDARY OUTCOMES:
Evolution of EBOV semen RNA and infectious loads | Semen collection will be performed at least at Day 7, Day 14, Day 21 and Day 90
  From Day 14 to Day 90, semen EBOV PCR will be performed every 3 weeks until their semen tests negative for virus twice by RT-PCR, with an interval of one week between tests.
Plasma and semen trough concentrations of favipiravir | Plasma collection at Day 3, Day7, Day 10 and Day 14. Semen collection at Day 7 and Day 14
Genetic variations associated with favipiravir exposition | Blood collection at Day 1 will be used for further genotyping.

CONTACTS AND LOCATIONS:
Overall Officials: Daouda Sissoko, Doctor, Principal Investigator — Inserm 897 unit, ISPED, Université de Bordeaux, Bordeaux cedex
Locations (2):
- Guinea (2):
  - Conakry, Conakry
  - Nzérékoré, Nzérékoré

REFERENCES:
- [Result] Eloy P, Laouenan C, Beavogui AH, Keita S, Manchon P, Etard JF, Sissoko D, Mentre F, Malvy D. High doses of favipiravir in two men survivors of Ebola virus disease carrying Ebola virus in semen in Guinea. IDCases. 2022 Jan 21;27:e01412. doi: 10.1016/j.idcr.2022.e01412. eCollection 2022. PMID 35127447